CLINICAL TRIAL: NCT07361575
Title: A Single-blind, Randomized Study Comparing the Quality of Colon Cleanliness With Prepackaged LRD (Low-residue Diet) vs. Guided (POG).
Brief Title: Study Comparing the Quality of Colon Cleanliness With Prepackaged LRD (Low-residue Diet) vs. Guided (POG).
Acronym: POG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Paris-Bercy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: POG
Record Dates: First submitted 2025-12-03; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer Prevention; Colorectal Cancer (Diagnosis); Colorectal Adenocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Disease | interventions — Colonoscopy; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with LRD prepared 24 hours before colonoscopy (Experimental): The LRD prepared is Colobox
  Interventions: Procedure: Colonoscopy; Other: Questionnaires; Other: Pre-colonoscopy diet
- Patients with not prepared LRD, 24 hours before colonoscopy (Active Comparator): The LRD is only explained orally and in writing to the patient
  Interventions: Procedure: Colonoscopy; Other: Questionnaires; Other: Pre-colonoscopy diet

INTERVENTIONS:
Procedure: Colonoscopy — Colonoscopy performed and Boston score evaluated
Other: Questionnaires — LRD satisfaction questionnaire LRD compliance questionnaire
Other: Pre-colonoscopy diet — 24 hours before the colonoscopy, The patients follow a special diet, either by themselves according to the investigator's oral instructions or by following a special preparation, Colobox.

SUMMARY:
Low-residue diet (LRD) in patient improves the quality of the colon cleanliness and thus the adenoma detection rate (ADR). This is a key criterion in colonoscopy screening for colorectal cancer (CRC). The benefit of an LRD lasting more than 24 hours before colonoscopy has not been demonstrated compared to a 24-hour LRD.

Few studies have evaluated the benefit of a prepackaged 24-hour LRD compared to simply receiving oral and written LRD instructions during a consultation.

The aim of the study is to evaluate the usefulness of a prepackaged LRD (Colobox®) compared to simple LRD instructions on colon cleanliness (Boston score) in patients examined by endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patient of one of the investigators for total colonoscopy (no prior colonic surgery);
* Patient aged 18 years or older;
* Patient classified as ASA 1, ASA 2, or ASA 3;
* Not participating in any other current clinical trial;
* Free, informed, and signed consent;
* Patient affiliated with or a beneficiary of a social security scheme, according to Article L.1124-1 of the French Public Health Code;

Exclusion Criteria:

* Patient taking major psychotropic medications;
* Patient with uncontrolled diabetes;
* Patient with coagulation abnormalities preventing polypectomy: PT <50%, Platelets <50,000/mm³, current effective anticoagulation therapy (clopidogrel, prasugrel, or ticagrelor);
* Patient referred for removal of a known polyp;
* Chronic inflammatory bowel disease;
* Known colonic stenosis;
* Diverticulitis of less than 6 weeks duration;
* Pregnant, parturient, or breastfeeding woman;
* Patient deprived of liberty by administrative or judicial order, or under guardianship or limited legal protection;
* Patient unable to understand the objectives and constraints of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Boston Score | 1 day
  A 9-point system, helps them see how clean a patient's large intestine is during a colonoscopy. This scale divides the large intestine into three parts: right, middle, and left.
  Each part can score from :
  BBPS = 0 (per segment) : unprepared colon segment with mucosa not seen because of solid stool that cannot be cleared.
  BPPS=3 (per segment) : entire mucosa of the colon segment seen well, with no residual staining, small fragments of stool, or opaque liquid.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Paris Bercy, Charenton-le-Pont, France